CLINICAL TRIAL: NCT06471556
Title: Efficacy of Methylprednisolone Pulses in Neuroendocrine Celles Hyperplasia of Infancy : An Early Phase Study
Acronym: CORTICONEHI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230821; 2023-508132-65-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Cell Hyperplasia of Infancy
Keywords: neuroendocrine cells hyperplasia of infancy (NEHI); Persistent tachypnoea of infancy (PTI); Childhood interstitial lung diseases (chILD); IV Corticosteroids pulses; Methylprednisolone; Oxygen therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV Methylprednisolone pulses (Experimental)
  Interventions: Drug: IV Methylprednisolone pulses

INTERVENTIONS:
Drug: IV Methylprednisolone pulses — Six (6) pulses (max) are performed at a 4 weeks interval (+/- 10 days). Each pulse is a 3-days-6h-perfusions of Methylprednisolone (500mg and 120mg) 10mg/kg/day diluted in 50ml of saline under supervision of SpO2, heart rate, blood pressure /

SUMMARY:
Childhood interstitial lung diseases (chILD) are a heterogeneous group of rare and severe disorders with an estimated prevalence of 1/100,000. Among them, neuroendocrine cells hyperplasia of infancy (NEHI), also called persistent tachypnoea of infancy (PTI), is one of the most common aetiology (up to 16% of the cases). NEHI involves young infants (median age at onset 3 to 6 months) with tachypnoea, hypoxemia, crackles, retractions, failure to thrive and specific localizations of ground glass opacities (GGO) on chest CT-scan (paramediastinal areas and anterior lobes (right middle lobe and lingula). At diagnosis, most patients (50 to 100%) require oxygen supplementation that usually lasts for months to years, sometimes associated with nutritional support with eventual enteral nutrition. NEHI is believed to be related to an increased number of neuroendocrine cells in airway epithelial area. These cells are abundant in foetal life, when they play a role in regulating the lung development and decrease before birth.

There is no specific treatment for NEHI. The main treatment of chILD is corticosteroids. However, in NEHI, their efficacy is matter of debate. There is only a few NEHI cases series or cohorts all over the world, accounting for a maximum of 500 reported cases within only retrospective studies. Among them, United States and Argentina teams report supportive care only (oxygen therapy and nutritional support) whereas other teams, like the French ones largely uses IV corticosteroid pulses.

Unlike the majority of chILD, NEHI prognosis is usually good. However, at school-age, 26% of the patients remain symptomatic or have an abnormal lung function. Moreover, oxygen therapy significantly affects quality of life (QoL) of the children with ILD (-10.43/100 points, p=0.02) but also QoL and mood of their parents (unpublished data).

The present study hypothesis that corticosteroids are associated with a reduction of the length of oxygen support in infants with NEHI.

DETAILED DESCRIPTION:
This study aims at assessing the beneficial effect of IV methylprednisolone pulses on oxygen therapy in infants with NEHI. It applies to all hypoxic NEHI patients aged below 12 months and followed in one of the centres of the RespiRare network. 18 patients will be recruited.

CORTICO-NEHI is designed as an early phase study following an A'Hern's Single Stage Phase II design.

All the patients are included in a single group receiving as a standard of care a maximum of 6 IV pulses of 3 days each.

12 visits will be performed as a standard of care:

* Screening visit (M-1 at maximum) :follow-up routine visit, (usually the hospitalization for NEHI diagnosis). If the patient is eligible, parents are informed of the study and an informed note is given. Information on the study protocol is given to obtain their written consent as soon as possible, and at the latest at the inclusion.
* Inclusion (M0) : After checking of the inclusion criteria and the absence of exclusion criteria, information and collection of parental consent. Following these investigations, the patient's first IV methylprednisolone pulse (D1) is administrated within the limit of 10 days.
* Treatment visits (M0 - M5): During a hospitalization, 6 pulses are performed at a 4 weeks interval (+/- 10 days). Each pulse is a 3-days-6h-perfusions of Methylprednisolone (500mg and 120mg) 10mg/kg/day diluted in 50ml of saline under supervision of SpO2, heart rate, blood pressure / 30min. If oxygen can be stopped (2 oxymetries with a 1-week interval +/- 10 days): The endpoint is reached and the methylprednisolone pulses are definitively stopped.
* Follow-up visits (M6, M9, M12, M15 and M18)

For the research needs,

* CT scan and Echocardiography will be done at inclusion if not performed in the past 3 months
* QoL questionnaires will be performed at inclusion, M6, M12 and M18
* Dipstick for sugar will be performed at M6, M9, M12, M15, M18 (in addition to M0 - M5 according to the standard of care)

ELIGIBILITY:
Inclusion Criteria:

* Infant aged under 12 months
* NEHI diagnosis based on:

  * The recently validated clinical Liptzin score ≥7/10 associated with a suggestive thoracic CT pattern with ground glass opacities confined to middle lobe, lingula, and paramediastinal lung areas OR
  * a clinical and thoracic CT suspicion and a lung biopsy showing an increased number of neuroendocrine cells in the epithelial airways area (at least one bronchiole with at least 10% of neuroendocrine cells)
* Oxygen requirement (awake and/or asleep) based on the usual pediatric recommendations (see section 4.1.1)
* Followed in one of the RespiRare participating centers
* Written informed consent of the holder(s) of its legal representative at the inclusion

Exclusion Criteria:

* Other cause of chILD assessed by lab biology tests, genetic analysis for surfactant genes (if available), bronchoalveolar lavage, and/or lung biopsy.
* Patient treated with IV methylprednisolone pulses before (any time)
* Diabetes
* Uncontrolled arterial hypertension
* Absence of Health care insurance
* Ongoing infection
* Immunization with a live attenuated vaccine within the past two weeks
* Long term treatment with Azithromycin and/or Hydroxychloroquine
* Patients already included in an interventional study (RIPH1, clinical investigation or clinical trial)

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of children still requiring oxygen therapy | Month 18
  To evaluate the efficacy on oxygen therapy need of a 6 months methylprednisolone pulses in NEHI patients at M18.

SECONDARY OUTCOMES:
Time to achieve the oxygen therapy weaning | Month 18
  Duration between randomization and the absence of oxygen therapy requirement at M18
The number of patients requiring continuous oxygen therapy (meaning sleep and awake oxygen therapy by opposition to sleep oxygen only) over time | Month 18
  Number of children still requiring oxygen therapy/ Number of children requiring only sleep oxygen
The number of patients requiring only sleep oxygen over time | Month 18
  Number of children requiring only sleep oxygen
The number of patients with a normal respiratory rate | Month 18
  Number of children with a normal respiratory rate at rest
ChILD healing (reduction of severity) over time | Between Month 0 and Month 18
  Difference of Fan's severity score assessing the severity of children with ILD (respiratory symptoms, SpO2<90% at sleep or exertion, SpO2<90% at rest and pulmonary hypertension)
Parents QoL | Month 0 and Month 18
  Family impact PedsQL score and a parents QoL score (submitted for publication)
Patient's QoL | Month 0 and Month 18
  Patients impact PedsQL and the chILD QoL scores; the chILDPQoL score.
Impact of NEHI on feeding and growth status | Between Month 0 and Month 18
  Number of patients requiring at least one enteral nutrition episode (based on the physician appreciation in case of abnormal weight curve)
Safety of methylprednisolone pulses | Between Month 0 and Month 18
  Number of unexpected hospitalizations for a respiratory exacerbation
Number of antibiotic courses for an infectious lung exacerbation | Between Month 0 and Month 18
  Safety of methylprednisolone pulses
Safety of methylprednisolone pulses | At Month 6
  * the number of patients with at least once systolic or diastolic arterial blood pressure (AP) over 2SD for the age at the days of methylprednisolone pulses
  * the number of patients with at least one elevated fasting glycaemia before the first day of methylprednisolone pulses.
Safety of methylprednisolone pulses | At Month 6
  - the number of patients with at least one elevated fasting glycaemia before the first day of methylprednisolone pulses.
To compare the family impact PedsQL questionnaire to the newly described chILD-PQoL questionnaire | Month 0, Month 6, Month 12, Month 18
  Correlation between family impact PedsQL questionnaire and the newly described chILD-PQoL questionnaire
To study thoracic CT-scan evolution | at Month 6 and Month 18
  Number of patients with an extension, a stability, a decrease or an absence of the GGO lesions on the CT-scan

CONTACTS AND LOCATIONS:
Overall Officials: Nadia NATHAN, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pediatric Pulmonology Department and Reference centre for rare lung diseases, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided